CLINICAL TRIAL: NCT05969743
Title: Letermovir Prophylaxis for CMV in Patients With Graft-versus-host Disease After Allogeneic Hematopoietic Cell Transplantation: a Proof of Concept Multicenter Study
Brief Title: Letermovir Prophylaxis for Cytomegalovirus (CMV) in Patients With Graft-versus-host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0827-22-RMC
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Graft-versus-host-disease; CMV
MeSH Terms: conditions — Graft vs Host Disease | interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Letermovir (Experimental): Patients meeting the inclusion criteria will receive letermovir 480 mg per day. Patients receiving concomitant cyclosporine will receive 240 mg of letermovir. Letermovir will be given during 14 weeks or until prednisone dose is reduced below 0.2 mg / kg / day, whichever comes earlier.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Patients meeting the inclusion criteria will receive letermovir 480 mg per day. Patients receiving concomitant cyclosporine will receive 240 mg of letermovir. Letermovir will be given during 14 weeks or until prednisone dose is reduced below 0.2 mg / kg / day, whichever comes earlier.

SUMMARY:
Explore the tolerability and efficacy of letermovir in the prevention of CMV reactivation in patients with acute and chronic graft-versus-host disease (GVHD) beyond day 100.

DETAILED DESCRIPTION:
42 patients meeting the inclusion criteria will receive letermovir 480 mg per day. Patients receiving concomitant cyclosporine will receive 240 mg of letermovir. Letermovir will be given during 14 weeks or until prednisone dose is reduced below 0.2 mg / kg / day, whichever comes earlier.

All the patients will continue herpesvirus prophylaxis with acyclovir or valacyclovir.

Patients will be evaluated biweekly until letermovir discontinuation. A PCR CMV test will be performed biweekly. Patients in whom clinically significant CMV infection (defined as CMV disease or CMV viremia leading to preemptive treatment) develop, will discontinue the trial regimen and begin anti-CMV therapy according to local practice. The threshold for preemptive treatment for CMV viremia will be >1000 copies/ ml.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* After allogeneic transplantation
* Seropositive for CMV
* Who already received letermovir prophylaxis until day 100 without CMV reactivation
* Beyond day 100 after transplantation at enrollment
* With acute or chronic GVHD
* Daily prednisone dose ≥ 0.5 mg/kg (or equivalent dose of another glucocorticoid) at enrollment.
* Negative polymerase chain reaction (PCR) for CMV at enrollment
* Provided informed consent

Exclusion Criteria:

* Seronegative for CMV
* Positive PCR for CMV at enrollment
* Patient has previously had CMV reactivation under letermovir.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of CMV infection | 14 weeks
  The proportion of patients with clinically significant CMV infection through week 14 after enrollment or until prednisone dose is reduced below 0.2 mg / kg / day, whichever comes earlier.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Yeshurun, MD, Principal Investigator — Institution of Hematology, Rabin Medical Center

IPD SHARING:
Plan to Share IPD: No